CLINICAL TRIAL: NCT04783545
Title: A Two-part, Double-blind, Placebo-controlled, Phase I Study of the Safety and Pharmacokinetics of Single and Multiple Ascending Doses of Intravenous VLX-1005 in Healthy Subjects
Brief Title: Phase I Study of VLX-1005 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Veralox Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VLX-1005-001
Record Dates: First submitted 2021-02-26; First posted 2021-03-05 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Safety and Tolerability in Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Single Ascending Dose Cohorts 1-6 (Experimental): Drug: VLX-1005
  Interventions: Drug: VLX-1005
- Single Ascending Dose Cohorts 1-6, Placebo (Placebo Comparator): Drug: Placebo
  Interventions: Drug: Placebo
- Multiple Ascending Dose Cohorts 7-9 (Experimental): Drug: VLX-1005
  Interventions: Drug: VLX-1005
- Multiple Ascending Dose Cohorts 7-9, Placebo (Placebo Comparator): Drug: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VLX-1005 — VLX-1005 infusion
  Arms: Multiple Ascending Dose Cohorts 7-9; Single Ascending Dose Cohorts 1-6
Drug: Placebo — Placebo infusion
  Arms: Multiple Ascending Dose Cohorts 7-9, Placebo; Single Ascending Dose Cohorts 1-6, Placebo

SUMMARY:
The principal objective of this study is to describe the safety of and tolerability to single and multiple doses of VLX-1005 in healthy subjects following intravenous (IV) administration.

Other exploratory objectives are:

To evaluate the pharmacokinetics and pharmacodynamics of VLX-1005 following IV administration.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, male or female (non-lactating and not of childbearing potential) subjects age 19 to 55 inclusive.
2. Females must have undergone one of the following sterilization procedures at least 6 months prior to the first dosing:

   1. hysteroscopic sterilization
   2. bilateral tubal ligation or bilateral salpingectomy
   3. hysterectomy
   4. bilateral oophorectomy; or be postmenopausal with amenorrhea for at least 1 year prior to the first dosing and follicle stimulating hormone (FSH) serum levels consistent with postmenopausal status.
3. Good general health, with no significant medical history. Subjects must have no clinically significant abnormalities on physical examination at screening, and/or before administration of the initial dose of study drug.
4. Body weight ≥ 50 kg at the screening visit.
5. Body Mass Index (BMI) between 18 and 32 kg/m2 inclusive.
6. Has laboratory values (clinical chemistry and hematology) within the normal reference range. Deviations from this range may be acceptable if they are considered 'not clinically significant' (NCS) by the PI.
7. Males who have not been vasectomized participating in the study must agree to use at least 2 approved methods of contraception (ie double-barrier or barrier plus hormonal), or abstain from sexual intercourse, from Day -2 to 4 weeks after dosing (or last dose Parts B)
8. Is a non-smoker and must not have used any nicotine products within three months prior to screening.
9. Able and willing to attend the necessary visits to the study center.

Exclusion Criteria:

1. Blood donation or recipient of blood transfusion in previous 12 weeks.
2. History of clinically significant endocrine, neurological, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases. Cardiovascular history should include assessment of risk factors for Torsades de Pointes Risk (e.g., heart failure, pulmonary edema, cardiomyopathy, hypokalemia, hypomagnesemia, or hypocalcemia, or family history of Long QT Syndrome, syncope or sudden death).
3. History of neoplastic disease (with the exception of adequately treated non-melanomatous skin carcinoma).
4. Mentally or legally incapacitated (e.g., has significant emotional problems at the time of Screening Visit or expected during the conduct of the study, or has a history of a clinically significant psychiatric disorder within the last 5 years).
5. Fever (body temperature >38C) or symptomatic viral/bacterial infection or use of antibi-otics within 2 weeks prior to Screening.
6. Supine resting blood pressure (BP) >140/90 mmHg or heart rate (HR) outside the range 40 to 100 beats per minute at Screening and at Day -1.
7. Clinically significant abnormality on ECG performed at the Screening Visit or prior to administration of the initial dose of study drug. (Sick sinus syndrome, second or third degree atrioventricular block, myocardial infarction, symptomatic or significant cardiac arrhythmia, prolonged QTcF interval, or bundle branch block.
8. Out of range (on repeat) testing for coagulation tests including fibrinogen.
9. Clinically significant laboratory abnormalities including: Impaired renal function (estimated creatinine clearance (CrCl) of <80 mL/minute based on CrCl = (140-age [years])(body weight [kg])/(72)(serum creatinine [mg/dL])).
10. Positive test for hepatitis C antibody, hepatitis B surface antigen, or human immunodefi-ciency virus (HIV) antibody at Screening.
11. Participants with a positive toxicology screening panel (urine test including qualitative identi¬fication of barbiturates, tetrahydrocannabinol, amphetamines, benzodiazepines, opiates, cocaine, cotinine and ethanol).
12. Participants with a history of substance abuse or dependency or history of recreational IV drug use (by self-declaration).
13. Participant has a suspected history of alcohol abuse in the 6 months prior to screening.
14. Use of NSAIDs, aspirin or aspirin-containing medications (and other medications affecting platelet function [for example cilostazol, clopidogrel, ticagrelor, prasugrel, dipyridamole]) in the 14 days prior to dosing with study medication.
15. Unable to refrain from or anticipates the use of any medications, including prescription and non-prescription drugs and herbal remedies (such as St. John's Wort [Hypericum perforatum]), beginning 14 days (or 5 half-lives, whichever is longer) before administration of the initial dose of study drug and continuing throughout the study until the final study visit. There may be certain medications that are permitted at the discretion of the Investigator and Sponsor (including paracetamol/acetaminophen, medications for the treatment of AEs following administration of study drug).
16. Subjects who are unlikely to comply with the study protocol or, in the opinion of the investigator, would not be a suitable candidate for participation in the study.
17. Have participated in any other investigational drug trial within 30 days of dosing in the present study.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2022-01-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants Reporting One or More Treatment-emergent Adverse Events | Baseline up to Day 29
Number of Participants Who Meet the Markedly Abnormal Criteria for Vital Sign Measurements at Least Once Post Dose | Baseline up to Day 29
Number of Participants Who Meet the Markedly Abnormal Criteria for 12-lead Electrocardiogram (ECG) or Telemetry Parameters at Least Once Post Dose | Baseline up to Day 29
Number of Participants Who Meet the Markedly Abnormal Criteria for Laboratory Values at Least Once Post Dose | Baseline up to Day 29

SECONDARY OUTCOMES:
AUC(inf) | day 1 pre-infusion and at multiple time points (up to 36 hours) post infusion
  Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for VLX-1005
C(max) | day 1 at the end of infusion (1 hour after infusion starts)
  Plasma Concentration at the end of Infusion for VLX-1005
T1/2 | day 1 pre-infusion and at multiple time points (up to 36 hours) post infusion
  Terminal Disposition Phase Half-life for VLX-1005
Pharmacodynamics of 12-Lipoxygenase Inhibition | day 1 pre-infusion and at multiple time points (up to 36 hours) post infusion
  12-HETE measurement in serum

CONTACTS AND LOCATIONS:
Overall Officials: Allen Hunt, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Inc., Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Undecided